CLINICAL TRIAL: NCT06212973
Title: A Phase 3, Multicenter, Randomized, Double-masked, Active Controlled Study to Evaluate the Efficacy and Safety of Epinastine Hydrochloride Eye Drops 0.05% in the Treatment of Chinese Seasonal Allergic Conjunctivitis Patients
Brief Title: A Study to Evaluate the Efficacy and Safety of Epinastine Hydrochloride Eye Drops in the Treatment of Chinese Seasonal Allergic Conjunctivitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZKO-EPI-202111
Record Dates: First submitted 2024-01-02; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Seasonal Allergic Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epinastine hydrochloride eye drops group (Experimental): Administered Epinastine hydrochloride eye drops+Simulating Azelastine hydrochloride eye drops bilaterally, twice daily
  Interventions: Drug: Epinastine Hcl Oph Soln+Simulating Azelastine Hcl Oph Soln
- Azelastine hydrochloride eye drops group (Active Comparator): Administered Azelastine hydrochloride eye drops+Simulating Epinastine hydrochloride eye drops bilaterally, twice daily
  Interventions: Drug: Azelastine Hcl Oph Sol+Simulating Epinastine Hcl Oph Soln

INTERVENTIONS:
Drug: Epinastine Hcl Oph Soln+Simulating Azelastine Hcl Oph Soln — Epinastine Hydrochloride Eye Drops + Simulating Azelastine Hydrochloride Eye Drops are used: both eyes are administered twice daily, once in the morning and once in the evening, with an interval of 8-12 hours between administrations; each time, 1 drop of each of the two eye drops is placed in each eye into the conjunctiva, and the two eye drops are applied at intervals of more than 5 minutes.
  Arms: Epinastine hydrochloride eye drops group
Drug: Azelastine Hcl Oph Sol+Simulating Epinastine Hcl Oph Soln — Azelastine Hydrochloride Eye Drops + Simulating Epinastine Hydrochloride Eye Drops are used: both eyes are administered twice daily, once in the morning and once in the evening, with an interval of 8-12 hours between administrations; each time, 1 drop of each of the two eye drops is placed in each eye into the conjunctiva, and the two eye drops are applied at intervals of more than 5 minutes.
  Arms: Azelastine hydrochloride eye drops group

SUMMARY:
The goal of this multicenter, randomized, double-blind, active control, non-inferiority clinical trial is to evaluate the efficacy of epinastine hydrochloride eye drops for the treatment of seasonal allergic conjunctivitis using azelastine hydrochloride eye drops as a positive control in Chinese patients. The main question it aims to answer are:

• Is the efficacy for of epinastine hydrochloride eye drops for the treatment of seasonal allergic conjunctivitis non-inferior to azelastine hydrochloride eye drops?Participants will be randomly assigned to the test group or control group in a 1:1 ratio. The test group was treated with epinastine hydrochloride eye drops + azelastine hydrochloride simulating eye drops, and the control group was treated with azelastine hydrochloride eye drops + epinastine hydrochloride simulating eye drops, which were used twice a day for 14 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign the informed consent form, and able to comply with the treatment plan, visits, and laboratory tests stipulated in the study. subjects under 18 years of age and without full capacity for civil behavior are required to sign the informed consent form in writing, and a legal guardian is also required to sign the informed consent form;
2. The age on the date of signing the informed consent is equal to or greater than 12 years old, gender is not limited;
3. Have any one of the following three laboratory report records prior to randomization:

   1. Positive eosinophil cytology results;
   2. Positive specific immunoglobulin E (IgE) test;
   3. Positive skin prick test;
4. Clinician-diagnosed seasonal allergic conjunctivitis in both eyes based on history, symptoms, and signs.

Exclusion Criteria:

1. Presence of ocular diseases that may affect the study results at the time of screening in either eye, such as blepharitis, blepharitis, dacryoadenitis, dacryocystitis, infectious conjunctivitis, keratitis, moderate-to-severe dry eye (according to the diagnostic grading of the Chinese expert consensus on dry eye), and uveitis;
2. Conjunctival inflammatory proliferative lesions (including giant papillary hyperplasia, paving stone-like hyperplasia, jelly-like hyperplasia, etc.) within 2 years prior to screening in either eye;
3. Best corrected visual acuity (BCVA) of less than 4.4 (five-point visual acuity) in either eye at screening;
4. Intraocular pressure>21 mmHg or <8 mmHg in either eye at screening;
5. Current or previous glaucoma or other optic nerve disease, or suspected glaucoma and other optic nerve disease, in either eye;
6. current or previous retinal detachment, diabetic retinopathy, or the presence of any progressive retinal disease in either eye;
7. Either eye has had internal eye surgery within 6 months prior to screening or has had laser eye surgery and external eye surgery within 3 months prior to screening or plans to have eye surgery during the study period;
8. Ocular trauma within 3 months prior to Screening in either eye (except where, in the judgment of the Investigator, there is no impact on the study validity and safety results);
9. Presence of a systemic disease at the time of screening that may affect the results of the study, e.g., dry syndrome, rheumatoid arthritis, graft-versus-host disease, systemic lupus erythematosus, scleroderma, and tuberculosis;
10. Presence of severe, unstable, or uncontrolled cardiovascular, cerebral, pulmonary, hepatic, renal, autoimmune, and other relevant systemic diseases at the time of screening, e.g., severe chronic obstructive pulmonary disease (COPD), severe asthma, severe cardiac arrhythmia, significant heart failure (New York Heart Association classification ≥ Class III), uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 90 mmHg ), uncontrolled diabetes, etc;
11. History of medical conditions that, in the judgment of the investigator, may interfere with the safe administration of topical antihistamines/mast cell stabilizers, such as hepatic or renal impairment (ALanine aminoTransferase(ALT) or ASpartate aminoTransferase(AST) ≥ 2.5 times the upper limit of normal; total bilirubin ≥ 1.5 times the upper limit of normal; and serum creatinine or urea/urea nitrogen ≥ 1.2 times the upper limit of normal), in the 6 months prior to screening;
12. The following topical (ophthalmic) prohibited drugs have been used or are planned to be used during the study period within the time period specified prior to randomization (the number of days is the pre-randomization period of prohibition and does not include experimental drugs):

    * Ocular immunosuppressive drugs (e.g. cyclosporine, tacrolimus, etc.): 60 days;
    * Ocular corticosteroid drugs (dexamethasone, flumethasone, prednisone acetate, rimexolone, difluprednate, loteprednol, etc.): 45 days;
    * Ocular mast cell stabilizing drugs: 14 days;
    * Ocular antihistamine and decongestant drugs: 3 days;
    * Ocular artificial tears: 1 day;
    * Other ophthalmic drugs: 3 days.
13. The following topical (dermal or nasal spray) prohibited medications have been used for the time specified prior to randomization or are planned to be used for the duration of the study (the number of days is the duration of prohibition prior to randomization):

    * Antihistamines and corticosteroids for periocular skin: 7 days;
    * Nasal spray immunosuppressive drugs: 60 days;
    * Nasal spray corticosteroid drugs: 45 days;
    * Nasal spray mast cell stabilizing drug: 14 days;
    * Nasal spray antihistamine and decongestant drugs: 3 days.
14. The following systemically prohibited drugs have been used or are planned to be used during the study period within the time period specified prior to randomization (the number of days is the time of prohibition prior to randomization):

    * Immunotherapy and immunosuppressive agents (including biologics): 60 days;
    * Long-acting corticosteroids (dexamethasone, betamethasone): 30 days;
    * Leukotriene receptor antagonists (e.g., montelukast sodium): 30 days;
    * Non-long-acting corticosteroids, mast cell stabilizers: 14 days;
    * Antihistamines, decongestants, monoamine oxidase inhibitors: 7 days;
    * Aspirin-containing drugs, non-steroidal anti-inflammatory drugs(NSAIDs): 3 days.
15. Non-pharmacological treatments to reduce the signs or symptoms of seasonal allergic conjunctivitis such as cold compresses to the eyes, desensitization therapy, and saline rinsing of the eyes are planned for the duration of the study;
16. Known allergic reaction to epinastine hydrochloride eye drops, azelastine hydrochloride eye drops, or any of the components of the simulated medications;
17. inability to avoid wearing contact lenses for the duration of the study;
18. participation in another clinical research trial within 30 days prior to randomization or planned during the study period;
19. women who are pregnant or breastfeeding; subjects who have a positive pregnancy test result at screening; do not consent to the use of an effective method of contraception from the start of the study until 4 weeks after the end of the study (including hormonal methods - oral, implanted, injectable, or transdermal birth control pills; physical barrier methods - - spermicide in combination with a physical barrier method such as a diaphragm or condom; an intrauterine device; or surgical sterilization of a partner, etc.) to avoid pregnancy in themselves or their partner within 4 weeks of study start to study end for subjects of childbearing age;
20. Presence of other factors that, in the opinion of the investigator, make participation in this study inappropriate, including inability or unwillingness to comply with the protocol (e.g., alcoholism, drug dependence, or psychological disorders, etc.).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline (Day 0) in independent investigator-rated ocular itch scores | Day 0~Day 14
  Changes from baseline (Day 0) in independent investigator-rated ocular itch scores were assessed at visit 5 (Day 14±2) (study eye). The ocular itch score was graded from 0 to 3(0=none, 1=mild, 2=moderate, 3=severe)

SECONDARY OUTCOMES:
Changes from baseline (Day 0) in independent investigator-rated total score of ocular itch, conjunctival hyperemia, and tearing total score | Day 0~Day 14
  Changes from baseline (Day 0) in independent investigator-rated total score of ocular itch, conjunctival hyperemia, and tearing total score at Visit 5 (Day 14±2)(study eye). The ocular itch score was graded from 0 to 3(0=none, 1=mild, 2=moderate, 3=severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No